CLINICAL TRIAL: NCT03224273
Title: Clinical Assessment of Two Inlay -Retained Bridge Designs (Proximal Box Shaped and Inlay Shaped) in Missing Posterior Teeth Cases
Brief Title: Clinical Assessment of Two Inlay -Retained Bridge Designs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Gomaa soliman, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-07-14
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Tooth Fractures
Keywords: proximal box design preparation
MeSH Terms: conditions — Tooth Fractures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ( proximal box design) (Experimental): The proximal box at least ( 1mm wide and has 6◦ divergences, and extend 2 mm apical to the isthmus ﬂoor.
  Interventions: Other: proximal box inlay retained bridge
- ( inlay shaped design) (Active Comparator): The occlusal inlay has a preparation depth of 2.0 mm for the ceramic. The occlusal preparation ( 4 mm wide and extend 4mm for premolar and 6 mm for molar mesiodistally
  Interventions: Other: proximal box inlay retained bridge

INTERVENTIONS:
Other: proximal box inlay retained bridge — inlay retained bridge is the less invasive type to restore single missing teeth in the posterior area
  Other Names: all ceramic inlay retained bridge

SUMMARY:
in the last years, dentistry is going to the concept of conservatism to preserve the most amount of tooth structure, so the evolution of new ceramic materials with invasive designs like (inlay- shaped and proximal box shaped) inlay retained bridge, the investigators can restore single missing posterior teeth with less invasive techniques and less rate of restoration fracture.

DETAILED DESCRIPTION:
It has been demonstrated that a great amount of tooth structure is lost during the prosthetic preparations of abutments for full-coverage FDPs with tooth substance removal of 63% of 73%, this aggressive loss of tooth structure usually accompanied with pain and postoperative sensitivity. In comparison With the inlay-retained bridge, there is less amount of tooth substance loss. this clinical study will provide benefits for practitioners and clinicians by guiding them to choose a more conservative treatment plan with the better marginal fit, clinical performance and satisfaction for the patients on the long term. rather than other benefits like less chair time, less risk for pulp injury, less time and cost

ELIGIBILITY:
Inclusion Criteria:

* Absence of periapical or periodontal or diseases
* sound abutment teeth or with small caries or filling on occlusal or proximal surfaces
* Maintenance of good oral hygiene
* No tooth mobility or grade 1 can be accepted
* Sufficient occluso-gingival tooth height (5mm)
* Good alignment of abutment teeth
* mesiodistal edentulous space preferred not exceed 12mm

Exclusion Criteria:

* Patients under the age of 18 or being incapable of taking out a contract
* Patients with any medical condition that impaired correct oral hygiene
* Endodontic ally treated abutment teeth
* a conspicuous medical or psychological history
* bruxism, or known allergic reaction to the materials used
* limited vertical space for the required connector height of 4mm
* pregnant female patients

Ages: 18 Years to 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
fracture | 1 year
  resistance of restoration to disintegrate and the assessment for the outcome will be done by using MUSPHS scale and the measuring unit is score